CLINICAL TRIAL: NCT01122888
Title: Pilot Biomarker Study of the Integrin AlphavBeta3 Antagonist Cilengitide (EMD121974) in Combination With Sunitinib
Brief Title: Cilengitide and Sunitinib Malate in Treating Patients With Advanced Solid Tumors or Glioblastoma Multiforme
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-01455; NCI-2011-01455 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000659080; UCCRC-09-259-A; 09-259-A (Other: University of Chicago Comprehensive Cancer Center); 8313 (Other: CTEP); P30CA014599 (NIH); U01CA069852 (NIH)
Record Dates: First submitted 2010-01-12; First posted 2010-05-13 (Estimated); Last update posted 2015-04-28 (Estimated); Status verified 2015-04

CONDITIONS: Adult Giant Cell Glioblastoma; Adult Glioblastoma; Adult Gliosarcoma; Adult Solid Neoplasm; Recurrent Adult Brain Neoplasm
MeSH Terms: conditions — Glioblastoma; Gliosarcoma; Brain Neoplasms | interventions — Cilengitide; Watchful Waiting

ARMS (2):
- Arm I (course 1) (Experimental): Patients receive cilengitide IV over 1 hour twice weekly for 2 weeks.
  Interventions: Drug: Cilengitide; Other: Laboratory Biomarker Analysis
- Arm II (course 1) (Other): Patients do not receive treatment and undergo a 2-week rest period.
  Interventions: Other: Clinical Observation; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Cilengitide — Given IV
  Other Names: EMD 121974; EMD-121974
  Arms: Arm I (course 1)
Other: Clinical Observation — Patients undergo a 2-week rest period
  Arms: Arm II (course 1)
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This clinical trial is studying how well giving cilengitide together with sunitinib malate works in treating patients with advanced solid tumors or glioblastoma multiforme. Cilengitide and sunitinib malate may stop the growth of tumor cells by blocking blood flow to the tumor. Giving cilengitide together with sunitinib malate may kill more tumor cells. Studying samples of blood in the laboratory from patients receiving cilengitide and sunitinib malate may help doctors understand the effect of these drugs on biomarkers.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the effect of cilengitide on changes in serum VEGFR2, a pharmacodynamic biomarker of sunitinib malate effects on endothelial function, during the withdrawal phase of a course of sunitinib malate in patients with advanced solid tumors or glioblastoma multiforme.

SECONDARY OBJECTIVES:

I. Determine the effect of cilengitide exposure on changes in VEGFR2 over the 14-day interval from the end of sunitinib malate administration to the end of course 1 in these patients.

II. Test the safety and efficacy of this regimen in these patients. III. Develop serum collagen c-telopeptide crosslinks (CTx) as a pharmacodynamic marker for cilengitide.

OUTLINE:

COURSE I: Patients receive oral sunitinib malate on days 1-14 (weeks 1-2). Patients are then randomized to 1 of 2 treatment arms.

ARM I: Patients receive cilengitide IV over 1 hour twice in weeks 3 and 4.

ARM II: Patients do not receive treatment in weeks 3 and 4.

COURSE II: Patients in both arms then receive oral sunitinib malate on days 1-14 and cilengitide IV over 1 hour twice in weeks 3 and 4. Treatment repeats every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up periodically.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed solid tumor or malignant glioblastoma multiforme meeting >= 1 of the following criteria:

  * Disease refractory to standard therapy
  * No standard therapy exists
  * Sunitinib malate monotherapy would be appropriate management
* Measurable disease is not required
* Previously treated brain metastases or primary brain neoplasms allowed provided patient is not receiving concurrent corticosteroids
* Karnofsky performance status 70-100%
* Absolute neutrophil count (ANC) >= 1,500/μL
* White blood cell count (WBC) >= 3,000/μL
* Platelet count >= 100,000/μL
* Hemoglobin >= 9 g/dL
* Total bilirubin normal (unless due to documented Gilbert syndrome)
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.5 times upper limit of normal (ULN) (< 5 times ULN in the presence of liver metastases)
* Creatinine normal OR creatinine clearance >= 60 mL/min
* Serum calcium =< 12.0 mg/dL
* QTc < 500 msec
* Patients with any of the following are allowed provided they have New York Heart Association (NYHA) class I-II cardiac function and undergo a baseline echocardiogram (ECHO)/multiple gated acquisition (MUGA):

  * History of class II heart failure and asymptomatic on treatment
  * Prior anthracycline exposure
  * Previously treated with central thoracic radiotherapy that included the heart in the radiotherapy port
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier contraception
* No history of allergic reactions attributed to compounds of similar chemical or biologic composition to sunitinib malate
* No concurrent uncontrolled illness including, but not limited to, any of the following:

  * Ongoing or active infection
  * Symptomatic congestive heart failure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * Psychiatric illness and/or social situation that would limit compliance with study requirements
* No pre-existing thyroid abnormality for which thyroid function cannot be maintained in the normal range with medication
* No documented thrombosis (pulmonary embolism or deep vein thrombosis) within the past 6 months
* No known coagulopathy or thrombophilia
* No proven gastric or duodenal ulcer or clinically significant gastrointestinal (GI) blood loss within the past 6 weeks
* No history of central nervous system (CNS) hemorrhage
* No life-threatening bleeding diathesis within the past 6 months
* No history of serious ventricular arrhythmia (i.e., ventricular fibrillation or ventricular tachycardia >= 3 beats in a row) or other significant electrocardiogram (ECG) abnormalities
* No poorly controlled hypertension (i.e., systolic blood pressure (BP) >= 150 mm Hg or diastolic BP >= 100 mm Hg)
* No condition that would impair the ability to swallow and retain sunitinib malate tablets, including any of the following:

  * GI tract disease resulting in an inability to take oral medications or a requirement for IV alimentation
  * Prior surgical procedures affecting absorption
  * Active peptic ulcer disease
* No gastrostomy, jejunostomy, or other forms of enteral tube feeding modalities
* None of the following conditions:

  * Serious or non-healing wound or ulcer
  * Abdominal fistula, GI perforation, or intra-abdominal abscess within the past 28 days
  * Cerebrovascular accident or transient ischemic attack within the past 12 months
  * Myocardial infarction, cardiac arrhythmia, stable/unstable angina, symptomatic congestive heart failure, or coronary/peripheral artery bypass graft or stenting within the past 12 months
  * NYHA class III or IV heart failure
  * Radiographically or physiologically diagnosed usual interstitial pneumonitis (UIP) or non-specific interstitial pneumonitis (NSIP)
* No bone fracture within the past 12 months
* No other concurrent anticancer agents or therapies
* More than 4 weeks since prior radiotherapy or systemic antineoplastic therapy (6 weeks for nitrosoureas, mitomycin C, or bevacizumab) and recovered
* More than 2 weeks since prior hormone replacement therapy or hormonal contraceptives
* More than 1 month since prior surgery
* At least 7 days since prior and no concurrent CYP3A4 inhibitors
* At least 12 days since prior and no concurrent CYP3A4 inducers
* Prior luteinizing hormone-releasing hormone agonists for hormone-refractory prostate cancer allowed
* Prior antiangiogenic agents (e.g., sorafenib, pazopanib, AZD2171 [cediranib maleate], PTK787 [vatalanib], or VEGF Trap [ziv-aflibercept]) allowed provided there is no disease progression
* No prior cilengitide or sunitinib malate
* No prior bevacizumab
* No other concurrent investigational agents
* No concurrent combination antiretroviral therapy for human immunodeficiency virus (HIV)-positive patients
* No concurrent agents with proarrhythmic potential (e.g., terfenadine, quinidine, procainamide, disopyramide, sotalol, probucol, bepridil, haloperidol, risperidone, indapamide, or flecainide)
* No concurrent palliative radiotherapy
* No other concurrent chemotherapy or biologic agents
* No concurrent medications that may cause QTc prolongation
* No concurrent therapeutic doses of coumarin-derivative anticoagulants (e.g., warfarin)

  * Up to 2 mg of daily warfarin for the prophylaxis of thrombosis allowed
  * Low-molecular weight heparin allowed provided prothrombin time (PT)/international normalized ratio (INR) =< 1.5
* No concurrent grapefruit juice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2009-12; Primary Completion 2012-09 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change in serum VEGFR2 | Over 14 days from the end of sunitinib to the end of course 1

SECONDARY OUTCOMES:
Comparison of the change in serum VEGFR2 in courses 1 and 2 | Over 14 days
  Compared using a paired t-test.
Progression-free survival | Assessed up to 30 days after completion of study treatment
  Estimated using the Kaplan-Meier method. Summarized by type, grade, and attribution and compared using chi-squared tests or Fisher exact tests, as appropriate.
Response rate evaluated using RECIST criteria | Up to 30 days after completion of study treatment
  Summarized by type, grade, and attribution and compared using chi-squared tests or Fisher exact tests, as appropriate.
Serum type I collagen c-telopeptide crosslink measurements | Up to 30 days after completion of study treatment
Toxicity rates, graded using the NCI CTCAE version 4.0 | Up to 30 days after completion of study treatment
  Compared using chi-squared tests or Fisher exact tests, as appropriate.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Maitland, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States